CLINICAL TRIAL: NCT00285493
Title: Phase 1 Study of Antibiotic Treatment for Low Back Pain
Brief Title: Low Back Pain and Antibiotic Treatment
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Withdrawn: study halted prematurely, prior to enrollment of first participant
Sponsor: Loewenstein Hospital (Other)
Collaborators: Clalit Health Services (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 230859
Record Dates: First submitted 2006-02-01; First posted 2006-02-02 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2011-06

CONDITIONS: Low Back Pain
Keywords: low back pain
MeSH Terms: conditions — Low Back Pain | interventions — Anti-Bacterial Agents

INTERVENTIONS:
Drug: Antibiotics

SUMMARY:
Clinical trial using antibiotic treatment, namely Rulid, after onset of low back pain.

DETAILED DESCRIPTION:
Clinical trial using antibiotic treatment, namely Rulid, after onset of low back pain.

ELIGIBILITY:
Inclusion Criteria:

- Must be able to swallow tablets

Exclusion Criteria:

- Allergy to antibiotics

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-01; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
protocol designed to assess or examine persons or groups in a systematic way to identify specific markers for eligibility for further evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Bambi Alyagon, MSc, Study Director — Loewenstein Hospital; Shoshana Weiler, MD, Principal Investigator — Loewenstein Hospital